CLINICAL TRIAL: NCT05319431
Title: An Open Label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of AK104 Plus Lenvatinib and TACE in the Treatment of Unresectable, Non-metastatic Hepatocellular Carcinoma
Brief Title: A Phase II Study of AK104 Plus Lenvatinib and TACE in HCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-216
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Unresectable, Non-metastatic Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK104+Lenvatinib+TACE (Experimental): Participants will receive AK104 IV every 3 weeks (Q3W) and Lenvatinib 12mg weight≥60kg or 8mg weight<60kg,PO QD The first Transarterial chemoembolization will be performed at the beginning of study.
  Interventions: Biological: AK104; Drug: Lenvatinib; Procedure: TACE

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 until disease progression or for a maximum of 24 months
Drug: Lenvatinib — Subjects will receive lenvatinib until disease progression or for a maximum of 24 months
Procedure: TACE — On demand TACE

SUMMARY:
To evaluate the efficacy and safety of AK104 plus lenvatinib combined with on-demand TACE in participants with unresectable, non-metastatic hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Histologically or cytologically documented hepatocellular carcinoma.
* CNLC IIa IIb or IIIa
* The main portal vein was not completely obstructed,
* Child-Pugh A or B
* At least one measurable lesion according to RECIST criteria
* ECOG PS 0-1
* Adequate organ function
* Estimated life expectancy of ≥3 months
* For women of childbearing potential: agreement to remain abstinent; For men: agreement to remain abstinent

Exclusion Criteria:

* Histologically or cytologically documented fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma, etc
* For HCC lesions ≥ 10 cm in any dimension, imaging evaluation showed that there were more than 10 lesions
* The main portal vein and the left and right primary branches were clogged with cancer thrombus
* History of hepatic encephalopathy or liver transplantation
* Any risk of bleeding; severe bleeding tendency or coagulation dysfunction, or under thrombolytic therapy.
* Occurred arteriovenous thromboembolic events within 6 months before the first administration.
* Inadequately controlled hypertension.
* Attack of symptomatic congestive heart failure (LVEF<50%); History of congenital long QT syndrome.
* Known presence or history of interstitial lung disease or required hormone treatment interstitial lung disease.
* Severe infections.
* Receipt of any anti-tumor treatment, chemotherapy, targeted therapy, immunotherapy,
* Enrollment of another clinical study within 4 weeks prior to the first administration of study drugs.
* Unable to receive an enhanced CT or MRI scan of the liver.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, which ever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR | Up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or PR, based on RECIST v1.1.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Number of participants with adverse events (AEs) | the time of informed consent signed through 90 days after the last dose
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Shao, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (5):
- China (5):
  - The First Hospital of Beijing University, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided